CLINICAL TRIAL: NCT00042354
Title: A Phase II, Open Label Study of Clofarabine in Pediatric Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Brief Title: Phase II Study of Clofarabine in Pediatric Acute Myelogenous Leukemia (AML) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO222
Record Dates: First submitted 2002-07-26; First posted 2002-08-01 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia, Myelocytic, Acute, Pediatric
Keywords: CLO222; clolar; Pediatric Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia | interventions — Clofarabine; Dosage Forms

INTERVENTIONS:
Drug: clofarabine (IV formulation)

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

The purpose of this study is to determine whether Clofarabine is safe and effective in the treatment of Acute Myelogenous Leukemia (AML.)

DETAILED DESCRIPTION:
This is a non-randomized, open label, Phase II study of Clofarabine in pediatric patients with refractory or relapsed acute myelogenous leukemia (AML). Eligible patients must be in first or subsequent relapse or be refractory. Forty eligible patients will be enrolled in a Fleming 2-stage sequential study design in order to better assess the efficacy and safety of clofarabine in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AML according to FAB classification with greater than or equal to 25% blasts in the bone marrow.
* Be less than or equal to 21 years old at time of initial diagnosis.
* Not be eligible for therapy of higher curative potential, and must be in first or subsequent relapse and/or refractory. Where an alternative therapy has been shown to prolong survival in an analogous population, this should be offered to the patient prior to discussing this study.
* Patients with acute promyelocytic leukemia (M3) must have been treated with at least 2 regimens-a retinoic acid-containing regimen and an arsenic trioxide-containing regimen before being considered for this study.
* Have a Karnofsky Performance Status (KPS) of greater than or equal to 70.
* Provide signed, written informed consent from parent or guardian and assent from patients greater than or equal to 7 years old according to local IRB and institutional requirements.
* Have adequate organ function as indicated by the following laboratory values, obtained within 2 weeks prior to registration: Serum bilirubin less than or equal to 1.5 x ULN; AST and ALT less than or equal to 5 x ULN; Serum Creatinine less than 2 x ULN for age. ULN= Institutional Upper Limit of Normal

Exclusion Criteria:

* Received previous treatment with Clofarabine.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Are pregnant or lactating. Male and female patients who are fertile must agree to use an effective means of birth control (i.e., latex condom, diaphragm, cervical cap, etc) to avoid pregnancy.
* Have psychiatric disorders that would interfere with consent, study participation, or follow up.
* Are receiving any other chemotherapy. Patients must have been off previous therapy for at least 2 weeks (with the exception of intrathecal therapy, which is allowed up to 24hrs prior to 1st dose of study drug) and must have recovered from acute toxicity of all previous therapy prior to enrollment. Treatment may start earlier, following consultation with the ILEX Medical Monitor, if there is evidence of disease relapse prior to that time.
* Have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Have symptomatic CNS involvement.
* Febrile neutropenia at time of study entry.
* Known or suspected fungal infection (ie. patients on parenteral antifungal therapy).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2002-05; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (18):
- United States (18):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital, Los Angeles, California
  - Children's Hospital, Orange County, California
  - Children's Hospital, San Diego, California
  - Children's Hospital, Denver, Colorado
  - University of Connecticut Health Center, Hartford, Connecticut
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering, New York, New York
  - Children's Hospital, Philadelphia, Pennsylvania
  - Children's Hospital, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Cook's Children's Medical Center, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas